CLINICAL TRIAL: NCT04093973
Title: Bicycle Exercise Echocardiography to Assess Physiological Significance of Mitral Annular Calcification
Status: Completed | Type: Observational
Sponsor: Albert Einstein Healthcare Network (Other)
Collaborators: Lantheus Medical Imaging (Industry)
Responsible Party: Principal Investigator, Gregg Pressman, Principal Investigator, Albert Einstein Healthcare Network
Other Study IDs: HN:4649
Record Dates: First submitted 2019-05-17; First posted 2019-09-18 (Actual); Last update posted 2023-05-24 (Actual); Status verified 2023-05

CONDITIONS: Mitral Annulus Calcification

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

GROUPS / COHORTS (2):
- MAC subjects: Outpatients with moderate to severe mitral annular calcification on echocardiogram who are able to perform supine bicycle exercise.
  Interventions: Diagnostic Test: bicycle stress echocardiography
- Controls: Sex matched individuals who are within 5 years of age of the paired MAC subject and who have the same left ventricular wall thickness as measured by echocardiography.
  Interventions: Diagnostic Test: bicycle stress echocardiography

INTERVENTIONS:
Diagnostic Test: bicycle stress echocardiography — Study subjects will perform supine bicycle exercise with echocardiography performed before, during, and after exercise. Definity (perflutren microbubble contrast agent) will be used as needed to enhance echo images.

SUMMARY:
Many people develop calcium deposits in the heart as they get older. One of the common places for this to occur is the mitral annulus, the band of tissue that supports the mitral valve (one of four heart valves). The purpose of this study is to examine effects of these deposits (termed mitral annular calcification or "MAC") on a person's ability to perform exercise. The research team will use ultrasound of the heart (Doppler echocardiography) to study people with MAC while they exercise on a specially designed bicycle.

DETAILED DESCRIPTION:
Mitral annular calcification (MAC) involves build-up of calcium in the mitral annulus, the fibro-muscular band which supports the mitral valve. The annulus aids in valve function, contracting in early systole (contraction phase) and bringing the valve leaflets together. In diastole (filling phase) it enlarges allowing blood to flow freely across the valve. Calcification stiffens the annulus and can extend onto the valve leaflets stiffening them. When severe, MAC impairs flow across the valve (mitral stenosis). This is characterized by a pressure gradient across the valve which can be detected by Doppler echocardiography (ultrasound).

Routine Doppler echocardiography is performed at rest when heart rates and flow across the mitral valve are low. Thus, even with severe MAC, there may only be a small pressure gradient present. However, with exercise these gradients can rise rapidly, leading to symptoms such as fatigue and shortness of breath.

MAC is associated with aging and is becoming more prevalent. Our hypothesis is that MAC is a common cause of shortness of breath with exertion. Further, the investigator believes this is under-appreciated because routine Doppler echocardiograms are done at rest. Therefore, the investigator will study adult subjects with moderate to severe MAC during bicycle exercise. Doppler echocardiography will be used to measure both the resting gradient across the mitral valve and changes with exercise. Symptoms will be measured by Borg Perceived Exertion scale.

If the research team is successful, the research team expects to demonstrate convincingly that this commonly encountered finding on Doppler echocardiography is an important cause of patient symptoms.

ELIGIBILITY:
Inclusion Criteria:

* At least moderate mitral annular calcification as judged by a previously published semi-quantitative echocardiographic score
* Over 18 years of age
* Able to use the semi-supine exercise bicycle
* Should be able to give informed consent.

Exclusion Criteria:

* Oxygen dependent lung or cardiac disease
* Moderate or greater aortic valvular disease
* Moderate or greater mitral regurgitation
* Reduced left ventricular ejection fraction, <35%
* Any diagnosed coronary disease
* A resting mean gradient of ≥10 mmHg across the mitral valve.

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: No vulnerable or special populations will be recruited for this study. In particular, those unable to or unwilling to consent, not yet adults, pregnant women and prisoners will be excluded.
Sampling Method: Non-Probability Sample
Enrollment: 40 (Actual)
Dates: Start 2014-11-07 (Actual); Primary Completion 2022-06-30 (Actual); Study Completion 2022-06-30 (Actual)

PRIMARY OUTCOMES:
Change in mean mitral valve gradient from baseline to peak exercise in patients with Mitral Annular Calcification compared to controls. | Procedure day
  Measuring how the pressure gradient across the mitral valve changes during exercise, and comparing these changes between subjects and controls.

SECONDARY OUTCOMES:
Change in pulmonary artery systolic pressure from baseline to peak exercise in patients with Mitral Annular Calcification compared to controls. | Procedure day
  Measuring how the blood pressure in the lungs changes during exercise, and comparing these changes between subjects and controls.
Borg Perceived Exertion Score at peak exercise in patients with Mitral Annular Calcification compared to controls. | Procedure day
  Comparing perceived exertion during exercise between subjects and controls. The Borg Scale of Perceived Exertion takes into account an individual's fitness level: It matches how hard a subject feels he/she is working, using numbers from 6 to 20; thus, it is a "relative" scale. The scale starts with "no feeling of exertion," which rates a 6, and ends with "very, very hard," which rates a 20. Moderate activities register 11 to 14 on the Borg scale ("fairly light" to "somewhat hard"), while vigorous activities usually rate a 15 or higher ("hard" to "very, very hard").

CONTACTS AND LOCATIONS:
Overall Officials: Gregg S Pressman, MD, Principal Investigator — Albert Einstein Healthcare Network
Locations (1):
- Einstein Medical Center, Philadelphia, Pennsylvania, United States

IPD SHARING:
Plan to Share IPD: No